CLINICAL TRIAL: NCT07308223
Title: 4th Affiliated Hospital, School of Medicine, Zhejiang University, China
Brief Title: Development of a Cloud-Based PRO (Patient-Reported Outcome) Management Program for Home-Based Cancer Pain Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KY-2025-047
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cancer Pain
MeSH Terms: conditions — Cancer Pain | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group received conventional telephone follow-up. Specifically, at 1 week and 3 weeks after discharge, ward follow-up nurses who had undergone standardized training conducted the follow-up using a pre-established checklist. The telephone calls covered pain intensity, location, medication usage, and adverse drug reactions.
- Intervention Group (Experimental): Prior to discharge, a nurse instructed patients on using the cloud-based follow-up platform. Patients then reported outcomes weekly via the platform using the PROMIS-29 profile. The system automatically monitored this data against preset thresholds; any exceedance triggered an alert to the care team for immediate assessment. Based on the reported data, the system also pushed personalized education on pain management and medication. Follow-up calls provided further guidance, including on non-pharmacological techniques to complement analgesic therapy.
  Interventions: Other: Proactive monitoring and patient education

INTERVENTIONS:
Other: Proactive monitoring and patient education — The intervention featured proactive monitoring of PRO data with threshold-based alerts, coupled with personalized patient education via the cloud and follow-up calls, to enhance timely care and self-management.
  Arms: Intervention Group

SUMMARY:
This study aims to develop and pilot a cloud-based Patient-Reported Outcomes (PROs) management program for home-based cancer pain patients within a hospital setting. It is expected to serve as a reference for improving pain management in home-based cancer care and to provide insights for future related research as well as the broader application and dissemination of the program.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;

  * Pathologically confirmed diagnosis of cancer with concomitant pain requiring analgesic medication; ③ Alert and oriented, free of psychiatric disorders or cognitive impairment; ④ Adequate comprehension, essentially normal vision and hearing, and basic literacy; ⑤ Proficient in using a smartphone (patient or primary caregiver), willing to accept cloud-platform follow-up and participate throughout the study;

    ⑥ Informed consent and voluntary participation.

Exclusion Criteria:

① Presence of severe psychiatric disorders;

② Critically ill or debilitated patients with advanced-stage tumor who are unable to complete the study procedures.

Withdrawal Criteria:

* Voluntary withdrawal or failure to complete the entire study process;

  * Death during follow-up; ③ Occurrence of accidents or clinical deterioration rendering continued participation infeasible; ④ Request to withdraw for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
pain intensity | 1 month
  Use the Numerical Rating Scale (NRS) to assess pain intensity

SECONDARY OUTCOMES:
Medication adherence | 1 month
  Morisky questionnaire on medication adherence

CONTACTS AND LOCATIONS:
Overall Officials: Huafang Zhang, MSN, Study Director — 4th Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 4th Affiliated Hospital, School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No